CLINICAL TRIAL: NCT00632281
Title: Stereotactic Body Radiation Therapy for Tumors in the Thorax
Brief Title: Stereotactic Body Radiation Therapy (SBRT) for Lung Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 502-2005
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Results first posted 2012-02-20 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2010-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Prescription dose: 48 Gy or 60 Gy RT

SUMMARY:
The purpose of this research study is to determine if Stereotactic Body Radiation Therapy(SBRT) is a good way to treat tumors near the thorax. Stereotactic Body Radiation Therapy (SBRT) is a general term for a group of techniques that are designed to deliver radiation therapy in a way that damages normal tissues less than conventional radiotherapy. The two features that distinguish SBRT from conventional therapy are procedures that decrease errors in patient positioning and technology that results in a radiation dose distribution that conforms more tightly to the tumor target. Patients will receive either 48 Gy or 60 Gy fractions depending on the type of tumor. The majority of patients will be treated in 1 week, Monday through Friday, with Wednesday off.

DETAILED DESCRIPTION:
Stereotactic Body Radiotherapy (SBRT) for tumors in the thorax is a relatively new therapy in the United States, but has been used extensively in Japan for more than 10 years. This protocol seeks to enroll patients in three broad categories based on histology and clinical scenario: primary therapy for non-small-cell lung cancer (NSCLC), primary therapy to thoracic metastases, and retreatment of previously irradiated tumors or lung.

Primary lung tumors

Several studies have been published describing the utility of Stereotactic Body Radiotherapy (SBRT) for primary untreated lung tumors. In the United States, the most influential has been the experience of Robert Timmerman at the University of Indiana (7). They enrolled 37 patients in a dose escalation trial of SBRT for T1 N0 and T2 N0 patients with Non-small-cell lung cancer (NSCLC). The trial began with 24 Gy given in 3 fractions and escalated to 60 Gy given in 3 fractions. Dose limited toxicity (DLT) was defined as any grade 3 pulmonary, esophageal, cardiac, or pericardial toxicity, or any grade 4 toxicity that was ascribed to the protocol treatment using the Common Toxicity Criteria from the National Cancer Institute. The maximum tolerated dose (MTD) was defined at dose where less and 2 of 5 enrolled patients experienced DLT. The MTD was not determined by this trial as this criteria was not met in the enrolled patients. Of the 37 patients, 2 experienced Grade 3 toxicity. One patient experienced pneumonitis and other patient experienced hypoxemia. Both patients responded to therapy and made full recoveries. There were no long term complications reported from the treatment at a mean follow-up of 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in this protocol
* Patients of all ages are eligible
* All tumor types are eligible
* Patients with prior thoracic radiotherapy and/or surgery are eligible
* Tumor size ≤ 5 cm

Exclusion Criteria:

* The subject is eligible for surgical resection or prefers treatment on this protocol to surgical resection.
* Less than 1 year since original radiation to thorax for retreatment patients.
* More than 2 tumors requiring SBRT
* The patient cannot be positioned reproducibly due to pain or other factors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amdur, MD, Principal Investigator — University of Florida- Radiation Oncology
Locations (1):
- University of Florida Shands Cancer Center, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients Receiving SBRT to Thorax: 22 patients had Non-small-cell lung cancer (NSCLC), 6 had metastatic disease, and 6 had 2 lesions treated simultaneously.
Period: Overall Study
Arm/Group | All Patients Receiving SBRT to Thorax
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients Receiving SBRT to Thorax
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 72.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Disease Status
Description: 2-year local control (Percentage of tumors that did not recur at treated site 2 years after treatment), cause-specific survival (percentage of patients who had not died from disease under study in the 2 years since treatment), overall survival (percent of patients still alive at 2 years after treatment), and freedom from failure (percentage of patients in whom the disease treated had not progressed or recurred in the 2 years since treatment)
Time Frame: 2 yrs
Population: 44 lesions in 38 patients were treated with IMRT or 3D conformal beams on a prospective trial examining thoracic SBRT. Twenty-two of 32 primary lung cancer patients had biopsy-proven NSCLC (stage IA, 21 patients; stage IB, 11 patients). Six had metastatic disease. Six patients had 2 lesions treated simultaneously.
Measure: Number; unit: percentage of participants
Arm/Group | All Patients Receiving SBRT to the Thorax
Number analyzed (Participants) | 38
percentage of participants
  Rate of 2-year control | 84
  Cause specific survival rate | 78
  Overall Survival rate | 55
  Freedom from Failure rate | 54

2. Secondary Outcome: Toxicity ot the Thorax
Description: Toxicity is defined as adverse events described in the CTCAE (version 3). Acute toxicity refers to adverse events that occurred up until 3 months after treatment and "late" toxicity as those occurring 3 months or longer after the end of treatment. Below are the Rates of grade 2 acute toxicity, grade 3 acute toxicity, late grade 3 toxicity, and late grade 4 toxicity
Time Frame: up to 2 years, 9 months
Measure: Number; unit: percentage of participants
Arm/Group | All Patients Receiving SBRT to the Thorax
Number analyzed (Participants) | 38
percentage of participants
  grade 2 toxicity | 30
  grade 3 toxicity | 2
  late grade 2 toxicity | 32
  late grade 3 toxicity | 8

ADVERSE EVENTS:
Time Frame: 2 years, 9 months
Description: Adverse events were assessed every 3 weeks for 3 months and then every 3 months.
Arm/Group | All Patients Receiving SBRT to Thorax
Serious Adverse Events (participants affected / at risk) | 20/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Receiving SBRT to Thorax (N=38)
Grade 3 Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Grade 3 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (24)
Grade 3 FEV1 (Respiratory, thoracic and mediastinal disorders) | 17 (33)
Grade 4 FEV1 (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Grade 3 Vital Capacity (Respiratory, thoracic and mediastinal disorders) | 6 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Receiving SBRT to Thorax (N=38)
Grade 1 cough (Respiratory, thoracic and mediastinal disorders) | 23 (85)
Grade 2 Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Grade 1 Dermatitis (Skin and subcutaneous tissue disorders) | 21 (41)
Grade 2 Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Grade 1 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (77)
Grade 2 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (61)
Grade 1 Esophagitis (Gastrointestinal disorders) | 1 (1)
Grade 2 Esophagitis (Gastrointestinal disorders) | 4 (10)
Grade 1 Fatigue (Investigations) | 29 (133)
Grade 2 Fatigue (Investigations) | 13 (29)
Grade 1 FEV1 (Respiratory, thoracic and mediastinal disorders) | 8 (16)
Grade 2 FEV1 (Respiratory, thoracic and mediastinal disorders) | 7 (18)
Grade 1 Fever (Infections and infestations) | 1 (1)
Grade 1 Nausea (Gastrointestinal disorders) | 16 (22)
Grade 2 Nausea (Gastrointestinal disorders) | 1 (1)
Grade 1 Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (8)
Grade 1 Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (19)
Grade 2 Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Grade 1 Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 10 (22)
Grade 2 Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Grade 1 Vital Capacity (Respiratory, thoracic and mediastinal disorders) | 9 (16)
Grade 2 Vital Capacity (Respiratory, thoracic and mediastinal disorders) | 21 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes